CLINICAL TRIAL: NCT05978245
Title: Obtaining Reliable Linguistic and Cultural Validation of the Questionnaires Cargier Bruden Inventony (CBI) and Zarit-12, Translate From English for Use in France
Brief Title: Obtaining Reliable Linguistic and Cultural Validation of the Questionnaires Cargier Bruden Inventony (CBI) and Zarit-12
Acronym: VALI-CBIZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0027_MPR
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Physical Medicine and Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To validate the 2 questionnaires ZARIT-12 and CBI it is important to go through several stages:

1. translation stage : during this stage there will be a meeting of experts to Validate the test version in French by 4 Bilingual translators of the French and English mother tongue.
2. pilot stage : recruit a number of 30 neurological patients' caregivers, in order to validate the comprehension, thus obtaining the final version of the questionnaire.
3. Validation stage : the two questionnaires have been validated, in this stage there should be a recruitment of 264 participants for the CBI questionnaire and 120 participants for the ZARIT-12 questionnaire, and these 2 questionnaires will be deliver to the participant on the same day.

   * The first questionnary will have to be filled the day they get the questionnary (day 1).
   * The second one must be completed and sent fourteen days later (day 14).

DETAILED DESCRIPTION:
To validate the 2 questionnaires ZARIT-12 and CBI it is important to go through several stages:

1. translation stage : during this stage there will be a meeting of experts to Validate the test version in French by 4 Bilingual translators of the French and English mother tongue.
2. pilot stage : recruit a number of 30 neurological patients' caregivers, in order to validate the comprehension, thus obtaining the final version of the questionnaire.
3. Validation stage : the two questionnaires have been validated, in this stage there should be a recruitment of 264 participants for the CBI questionnaire and 120 participants for the ZARIT-12 questionnaire, and these 2 questionnaires will be deliver to the participant on day 1. The first questionnary will have to be filled on day 1 and the second one must be completed and sent fourteen days later (so on day 14)

ELIGIBILITY:
Inclusion Criteria:

* Caregivers (family or friend) of patients followed for a central neurological pathology (MS, BM, Parkinson's, stroke, congenital (Spina...)) or peripheral (ponytail, peripheral neuropathies)
* Adult caregivers (age ≥ 18 years), regardless of the patient's age
* Francophone caregivers (ability to read, write and understand French)
* Caregivers who did not object to the use of their data or the patient's data for research

Exclusion Criteria:

* - Professional caregivers
* caregivers of patients being cared for with a pathology other than neurological
* Minor caregivers (age ≤ 17 years)
* Caregivers with no or poor French language skills
* Caregivers who refused to participate in the research

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulted in the hospital wards included in the research and suffering from neurological pathology with the inclusion of caregivers of patients who have had a consultation.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
French-language linguistic and cultural validation of caregiver burden questionnaires (Zarit-12) in a population of neurological patients | two days (day one and day fourteen)
  ZARIT-12
French-language linguistic and cultural validation of caregiver burden questionnaires (CBI) in a population of neurological patients | two days (day one and day fourteen)
  CBI questionnaire

SECONDARY OUTCOMES:
Identifying populations at higher risk of burden (ZARIT-12) | two days (day one and day fourteen)
  ZARIT-12
Identifying populations at higher risk of burden (CBI) | two days (day one and day fourteen)
  CBI questionnaire
Identification of risk factors for caregiver's burden (ZARIT-12) | two days (day one and day fourteen)
  ZARIT-12
Identification of risk factors for caregiver's burden (CBI) | two days (day one and day fourteen)
  CBI questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Delafontaine, Saint-Denis, Seine Saint Denis, France